CLINICAL TRIAL: NCT02740127
Title: Prospective Randomized Clinical Trial to Evaluate the Use of Caudal Nerve Blocks in Adult Penile Prosthesis Surgery
Brief Title: Evaluate Use of Caudal Nerve Blocks in Adult Penile Prosthesis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014-0990; NCI-2016-00860 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Results first posted 2021-09-30 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Malignant Neoplasms of Male Genital Organs
Keywords: Malignant neoplasms of male genital organs; Adult Penile Prosthesis Surgery; Caudal nerve block; CNB; General anesthesia; GA; Ropivacaine; Naropin; Epinephrine; Decadron; Dexamethasone; Clonidine; Propofol; Diprivan
MeSH Terms: interventions — Ropivacaine; Epinephrine; Calcium Dobesilate; Dexamethasone; Clonidine; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Caudal Nerve Block + General Anesthesia Group (Experimental): Participants receive a caudal nerve block (CNB) prior to surgery and receive general anesthesia during surgery.
  Study staff calls participant about 3 days after surgery.
  Interventions: Procedure: Caudal Nerve Block (CNB); Drug: Ropivacaine; Drug: Epinephrine; Drug: Decadron; Drug: Clonidine; Drug: Propofol; Behavioral: Phone Call
- General Anesthesia Alone Group (Active Comparator): Participants receive general anesthesia (GA) during surgery without a caudal nerve block.
  Study staff calls participant about 3 days after surgery.
  Interventions: Drug: Propofol; Behavioral: Phone Call

INTERVENTIONS:
Procedure: Caudal Nerve Block (CNB) — General anesthesia given in the OR using Propofol titrated for induction. CNB given as bolus injection into the caudal canal in the operating room (OR) by attending anesthesiologist using 1% Ropivacaine (max 5mg/kg) + 1:400,000 Epinephrine + Decadron 10 mg + Clonidine 100 mcg.
  Arms: Caudal Nerve Block + General Anesthesia Group
Drug: Ropivacaine — Ropivacaine 1 % (max 5mg/kg) by bolus injection given by anesthesiologist in OR.
  Other Names: Naropin
  Arms: Caudal Nerve Block + General Anesthesia Group
Drug: Epinephrine — Epinephrine 1:400,000 by bolus injection given by anesthesiologist in OR.
  Arms: Caudal Nerve Block + General Anesthesia Group
Drug: Decadron — Decadron 10 mg by bolus injection given by anesthesiologist in OR.
  Other Names: Dexamethasone
  Arms: Caudal Nerve Block + General Anesthesia Group
Drug: Clonidine — Clonidine 100 mcg by bolus injection given by anesthesiologist in OR.
  Arms: Caudal Nerve Block + General Anesthesia Group
Drug: Propofol — General anesthesia given in the OR using Propofol titrated for induction.
  Other Names: Diprivan
Behavioral: Phone Call — Study staff calls participant about 3 days after surgery to ask about their pain, amount of pain drugs they have taken, and how satisfied they are with the type of anesthesia and pain control they received. This call should last about 5-10 minutes.

SUMMARY:
During penile prosthesis surgery, patients are given general anesthesia in combination with other pain drugs. A caudal nerve block (CNB) is a local anesthetic injected near the tailbone, in addition to general anesthesia, which can lower the need for pain drugs.

The goal of this clinical research study is to learn how effective CNBs are in patients who are having penile prosthesis surgery compared to patients who only have general anesthesia by studying how long you stay in the hospital and the level of pain you have after surgery.

This is an investigational study. The general anesthesia and CNB used in this study are FDA approved and commercially available. It is considered investigational to compare the effectiveness of CNBs in penile prosthesis surgery to general anesthesia alone. The study doctor can explain how the study drugs are designed to work.

Up to 104 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups and CNB Administration:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. You will have an equal chance of being assigned to either group.

* If you are assigned to Group 1, you will receive a CNB and general anesthesia during surgery.
* If you are assigned to Group 2, you will only receive general anesthesia during surgery.

You will not know to which group you have been assigned. The CNB will be given to you while you are under general anesthesia. To receive a CNB, a special needle is inserted at the lower part of the back (near the tailbone). A type of local anesthesia is then injected into the sac surrounding the spinal cord that contains the nerves related to the penis.

All participants will also receive general anesthesia as part of their standard care. You will also receive a separate consent form for the surgery that explains the procedure and its risks, including the risks for general anesthesia.

After Surgery Data Collection:

During the 24 hours after surgery, the study staff will ask you to rate your pain on a scale of 0-10. You will be asked to rate your pain about every 30 minutes while you are in the hospital, but you may be asked to rate your pain more often if needed. It should take less than 5 minutes each time to rate your pain. Depending on how you rate your pain, additional pain drugs may be given to you as part of your standard care.

If you are discharged from the hospital on the same day as your surgery or if you are discharged before a member of the staff can ask you to rate your pain, the study staff will call you within 24 hours after you have been discharged from the hospital. This call should last about 5-10 minutes.

The amount of pain drugs given to you before, during, and after surgery will also be recorded.

About 3 days after your surgery, the study staff will call you to ask about your pain, the amount of pain drugs you have taken, and how satisfied you are with the type of anesthesia and pain control you have received. This call should last about 5-10 minutes.

Length of Study:

Your participation in this study will be over after the phone call about 3 days after your surgery has been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that consent to participate.
2. Patients undergoing penile prosthesis surgery.
3. Patients that are male.
4. Patients that are 18 years of age or older.

Exclusion Criteria:

1. Patients on chronic pain medications (ie. Chronic = more than once every two days for greater than 2 weeks) excluding Aspirin, Acetaminophen and NSAIDs.
2. Patients with a BMI > 40.
3. Patients with chronic pain syndromes.
4. Patients with hypersensitivity to Ropivacaine/amide-type anesthetics.
5. Prior surgery of the sacrum.
6. Patients taking anti-coagulants or other blood thinning medications prior to surgery during the specified time frames: i) Low molecular weight heparin less than 36 hours prior to surgery. ii) Coumadin less than 5 days prior to surgery. iii) Plavix and NSAIDs less than 7 days prior to surgery.
7. Patients on any anti-seizure medications, such as gabapentin or Lyrica, specifically for chronic pain management less than 24 hours prior to surgery
8. Patients on Celebrex less than 24 hours prior to surgery
9. Patients taking more than 81 mg of Aspirin daily

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Bellard, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- General Anesthesia and Caudal Nerve Block: If the patient is randomized to Group I, the patient will receive general anesthesia using Propofol titrated for induction. The airway will be secured thereafter. The caudal block will be performed as a bolus injection into the caudal canal in the OR by the attending anesthesiologist using 1% Ropivacaine (max 5mg/kg) + 1:400,000 Epinephrine + Decadron 10mg + Clonidine 100mcg. Patients will be continuously monitored by ASA guidelines. Anesthesia will be maintained with Sevoflurane 1.3-2.5% or Desflurane 2.5-8.5%, oxygen, air, nitrous oxide and Fentanyl as needed. At the completion of surgery, reversal of muscle relaxant with Glycopyrrolate 0.2mg IV for each 1mg IV of Neostigmine (max 5mg) will be given as indicated.
- General Anesthesia Only: Patients in Group II will receive general anesthesia using Propofol titrated for induction. The airway will be secured thereafter. Anesthesia will be maintained with Sevoflurane 1.3-2.5% or Desflurane 2.5-8.5%, oxygen, air, nitrous oxide and fentanyl as needed. At the completion of surgery, reversal of muscle relaxant with Glycopyrrolate 0.2mg IV for each 1mg IV of neostigmine (max 5mg) will be given as indicated.
Period: Overall Study
Arm/Group | General Anesthesia and Caudal Nerve Block | General Anesthesia Only
Started | 24 | 28
Completed | 24 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Anesthesia and Caudal Nerve Block | General Anesthesia Only | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 14 | 18 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 28 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24 | 28 | 52

OUTCOME MEASURES:

1. Primary Outcome: Post-Operative Pain Medication Usage in Post Anesthesia Care Unit (PACU)
Description: Pain evaluated by the amount of intravenous and oral pain medicine administered in the first 24 hours post-operatively. Pain assessed using the numeric rating scale (NRS). The NRS is scored by numeric integers, 0 through 10, where 0 is no pain and 10 is the worst pain.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | General Anesthesia and Caudal Nerve Block | General Anesthesia Only
Number analyzed (Participants) | 24 | 28
mg | 13.0208 (11.6362) | 15.1786 (16.6022)

2. Secondary Outcome: Post-operative Pain the First 24hrs
Description: To determine whether the use of a CNB in patients undergoing penile prosthesis surgery results in decreased immediate postoperative pain in the first 24 hours after surgery compared with patients having only general anesthesia as determined by postop pain score. The mean, median and max pain will be assessed using the numeric rating scale (NRS). The NRS is scored by numeric integers, 0 through 10. The NRS will be used verbally. Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | General Anesthesia and Caudal Nerve Block | General Anesthesia Only
Number analyzed (Participants) | 24 | 28
score on a scale
  Min Pain within 24hrs | 1.1667 (130.77) | 0.9286 (1.3859)
  Median Pain within 24 hrs | 3.0833 (2.2778) | 3.7143 (1.8926)
  Max Pain within 24 hrs | 6.125 (2.6096) | 6.7857 (2.0612)

3. Secondary Outcome: Length of Hospital Stay
Description: To determine whether the use of a CNB in patients undergoing penile prosthesis surgery results in a decreased length of hospital stay compared with patients having only general anesthesia.
Time Frame: 32 Hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | General Anesthesia and Caudal Nerve Block | General Anesthesia Only
Number analyzed (Participants) | 24 | 28
Hours | 24.8424 (4.9821) | 24.9506 (2.4564)

ADVERSE EVENTS:
Time Frame: 3 days post surgery
Arm/Group | General Anesthesia and Caudal Nerve Block | General Anesthesia Only
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 0/24 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT02740127/Prot_SAP_000.pdf